CLINICAL TRIAL: NCT03131609
Title: Avoiding Bacterial Contamination of Clean Catch Urine Cultures in Ambulatory Patients in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: EBLEN Charities (Unknown); Forte Medical Ltd. (Unknown); Avadim Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Mary Lough, Clinical Assistant Professor, Stanford University
Other Study IDs: 33879
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Urinary Tract Infections; Bacteriuria; Urinalysis
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria | interventions — Urine Specimen Collection; FTX, spider toxin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Container + Castile-soap wipe: Sterile urine collection container and Castile-soap wipe given to patient to self-obtain a clean catch mid-stream urine specimen - Control group represents usual care in the Emergency Department.
  Interventions: Other: Container; Other: Castile-soap wipe
- B: Container + Silver impregnated wipe: Sterile urine collection container and silver-impregnated cloth-wipe given to patient to self-obtain a clean catch mid-stream urine specimen
  Interventions: Other: Container; Other: Silver Impregnated Wipe
- C: Funnel + Castile-soap wipe: Sterile urine collection funnel and Castile-soap wipe given to patient to self-obtain a clean catch mid-stream urine specimen
  Interventions: Other: Funnel; Other: Castile-soap wipe
- D: Funnel + Silver-impregnated wipe: Urine collection funnel and sliver impregnated cloth-wipe given to patient to self-obtain a clean catch mid-stream urine specimen
  Interventions: Other: Silver Impregnated Wipe; Other: Funnel

INTERVENTIONS:
Other: Container — Ambulatory patients in the Emergency Department who have a urine culture ordered by the physician receive one of four urine collection/hygiene options.
  Other Names: Standard container for urine collection
  Groups: A: Container + Castile-soap wipe; B: Container + Silver impregnated wipe
Other: Silver Impregnated Wipe — Ambulatory patients in the Emergency Department who have a urine culture ordered by the physician receive one of four urine collection/hygiene options.
  Other Names: Theraworx
  Groups: B: Container + Silver impregnated wipe; D: Funnel + Silver-impregnated wipe
Other: Funnel — Ambulatory patients in the Emergency Department who have a urine culture ordered by the physician receive one of four urine collection/hygiene options.
  Other Names: Peezy Mid-stream urine collection kit
  Groups: C: Funnel + Castile-soap wipe; D: Funnel + Silver-impregnated wipe
Other: Castile-soap wipe — Ambulatory patients in the Emergency Department who have a urine culture ordered by the physician receive one of four urine collection/hygiene options.
  Groups: A: Container + Castile-soap wipe; C: Funnel + Castile-soap wipe

SUMMARY:
The purpose of this study is to find the best cleaning and collection methods to obtain a 'non-contaminated' clean catch mid-stream urine sample to diagnose suspected urinary tract infection (UTI).

DETAILED DESCRIPTION:
BACKGROUND: Urinary tract infection (UTI) is a major public health issue resulting in more than 3-million visits to Emergency Departments in the United States each year. As part of the diagnostic work up, a sterile urine sample is requested for culture. The preferred urine specimen is a "Clean Catch Midstream Urine Sample". When patients are ambulatory and competent, this is a self-obtained specimen in a private bathroom. If the urine is not collected in a sterile manner the urine sample may be 'contaminated' by bacteria that originate from the skin or genital area, and not from the urinary tract. This is often described by the clinical laboratory as 'mixed growth bacteria'. A contaminated sample may lead to a false-positive urine culture result. In a non-contaminated urine specimen, only a single bacterial growth is identified as the source of the infection. Mixed bacterial flora with two or more microorganisms makes interpretation of the urine culture more difficult and prone to error. The American College of Pathologists has published results of national laboratory surveys on Urine Culture Contamination in 1998 and 2008 that document the scope of the problem.

SAMPLE: Adult ambulatory patients in the Emergency Department who have a suspected UTI and have a urine culture ordered by a physician. A total of 2000 patients will be enrolled (500 per group). This is estimated to result in 600 urine samples (150 per group). Written consent is not normally required for a self-obtained urine sample. The study will be explained and participants will verbally consent or decline to participate, as approved by the Institutional Review Board.

SETTING: Emergency Department of an academic medical center.

METHOD: This is a randomized controlled trial (RCT) with 4 groups that compare different patient self-cleaning and self-collection methods. All study supplies materials are commercially available in the United States. Each participant will be provided with study-specific visual aids for male or female participants and their randomly assigned group. The four groups are:

Group 1: Standard moist wipes and standard collection container. Group 2: Silver impregnated moist wipes and standard collection container. Group 3: Standard moist wipes and funnel collection container. Group 4: Silver impregnated moist wipes and funnel collection container. The urine samples will be sent to the Hospital Microbiology Laboratory for analysis. Urine samples with a positive leuk-esterase pre-screen will be sent for urine culture.

DATA ANALYSIS:This study is powered to detect a large effect size change in any study groups (2. 3. 4) compared with control (group 1). The sample size is sufficient to identify the method(s) with the lowest urine sample contamination rate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of older
* Urine culture order by physician

Exclusion Criteria:

* Under 18 years of age
* Urinary catheter in place
* Not ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients in the Emergency Department at an Academic Medical Center with a physician order for a urine culture. Patient must be able to self-obtain the urine culture.
Sampling Method: Probability Sample
Enrollment: 1471 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Decrease in the number of contaminated urine cultures | 9 months
  Contamination >10,000 CFU/mL mixed flora identified by Clinical Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Lough, PhD, RN, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lough ME, Shradar E, Hsieh C, Hedlin H. Contamination in Adult Midstream Clean-Catch Urine Cultures in the Emergency Department: A Randomized Controlled Trial. J Emerg Nurs. 2019 Sep;45(5):488-501. doi: 10.1016/j.jen.2019.06.001. PMID 31445626